CLINICAL TRIAL: NCT04782037
Title: Effectiveness of Folic Acid Supplementation in Acute Watery Diarrhea Among Children Under 5 Years of Age
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: King Edward Medical University (Other)
Responsible Party: Principal Investigator, rafia Jamil, Post Graduate Resident (MD Pediatric Medicine), King Edward Medical University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 321/RC/KEMU
Record Dates: First submitted 2021-03-01; First posted 2021-03-04 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Diarrhoea;Acute
Keywords: acute watery diarrhea; folic acid; L-methylfolate

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- L-methylfolate supplementation (Experimental): Children under 1 year of age in group A will receive 3 drops (90mcg) of L-methylfolate calcium) while those older than 1 year of age will be given 5 drops (150mcg) daily fior 5 days
  Interventions: Drug: L-Methylfolate Calcium
- distilled water (Placebo Comparator): Subjects in Group B will receive equal amount of distilled water as placebo (i.e. 3 drops to <1yr age and 5 drops to >1 yr.
  Interventions: Drug: L-Methylfolate Calcium

INTERVENTIONS:
Drug: L-Methylfolate Calcium — Folic acid is one of the water-soluble B vitamins, which is synthetically-produced and found in fortified foods and supplements. It is essential for the synthesis and repair of DNA and RNA and metabolism of amino acids which are required for cell division. There is damage to the intestinal mucosa in most diarrhea cases; therefore, the role of folic acid has been studied as adjuvant therapy for diarrhea since folic acid plays an important role in the synthesis of DNA especially in rapidly regenerating cells.

SUMMARY:
Folic acid is a palatable and easily available drug with no serious adverse effects. L-methylfolate is its biologically activated form and is preferred because of its direct availability for certain metabolic processes. As there is no specific and safe drug available that may help in decreasing the duration of diarrhea, purging rate or consistency of stools; and having known the theoretical benefits of folic acid in this regard, it would be appropriate to assess the effectiveness of L-methylfolate among children with diarrhea.

DETAILED DESCRIPTION:
After approval from the Institutional Review Board of King Edward Medical University, Mayo Hospital, Lahore, all children diagnosed with acute watery diarrhea as per operational definition fulfilling the inclusion criteria, presenting to the Department of Pediatrics, Mayo Hospital, will be enrolled in this study.

Informed written consent will be taken from the parents/guardians of all participants. A detailed history and examination of each subject would be done by an investigator at presentation.

Patients will be randomized in two groups - A and B by lottery method. There will be 162 patients in each group. The treatment regimen that includes breast feeding, nutritional advice, rehydration plan; ORT by low osmolar ORS or intravenous rehydration (if required) and zinc sulphate will be given according to the WHO guidelines to all patients of both groups. Children under 1 year of age in group A will receive 3 drops (90mcg) of L-methylfolate calcium) while those older than 1 year of age will be given 5 drops (150mcg). Subjects in Group B will receive equal amount of distilled water as placebo (i.e. 3 drops to <1yr age and 5 drops to >1 yr. Frequency and grades of loose stools in both groups will be assessed daily and written down on a predesigned proforma.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 2months- 5 years
* Both genders
* Acute watery diarrhea as per operational definition
* Diarrhea of less than 7-day duration

Exclusion Criteria:

* Severely malnourished children <3 SD
* Bloody diarrhea
* Prolonged (7-14 days duration), persistent (>14 days duration) or chronic diarrhea (>4weeks duration)
* Those who received folic acid within the last 14 days
* Hospital-acquired diarrhea (diarrhea occurring after 48hrs of stay in hospital)
* Antibiotic-associated diarrhea.
* Presence of other co morbid conditions like pneumonia, sepsis, meningitis, etc.

Ages: 2 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 324 (Estimated)
Dates: Start 2020-10-21 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Changing the frequency of stools | 5 days
  L-methylfolate supplementation is effective in changing the frequency of stools. It will be measured in episodes per day
Effectiveness in improving grades of diarrhea | 5 days
  L-methylfolate supplementation is effective in changing grades of diarrhea. WHO grades will be taken as reference
Effectiveness in changing duration of diarrhea | 5 days
  L-methylfolate supplementation is effective in changing duration of diarrhea in days.

CONTACTS AND LOCATIONS:
Overall Officials: MUHAMMAD Haroon HAMID, MBBS,FCPS, Principal Investigator — CHAIRMAN PEDIATRIC MEDICINE, MAYO HOSPITAL; Sadia shabir, MBBS, FCPS, Principal Investigator — ASSISTANT PROFESSOR, PEDIATRIC MEDICINE UNIT 1, MAYO HOSPITAL
Locations (1):
- Mayo hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kotloff KL. The Burden and Etiology of Diarrheal Illness in Developing Countries. Pediatr Clin North Am. 2017 Aug;64(4):799-814. doi: 10.1016/j.pcl.2017.03.006. PMID 28734511
- [Background] GBD Diarrhoeal Diseases Collaborators. Estimates of global, regional, and national morbidity, mortality, and aetiologies of diarrhoeal diseases: a systematic analysis for the Global Burden of Disease Study 2015. Lancet Infect Dis. 2017 Sep;17(9):909-948. doi: 10.1016/S1473-3099(17)30276-1. Epub 2017 Jun 1. PMID 28579426
- [Background] Walker CLF, Rudan I, Liu L, Nair H, Theodoratou E, Bhutta ZA, O'Brien KL, Campbell H, Black RE. Global burden of childhood pneumonia and diarrhoea. Lancet. 2013 Apr 20;381(9875):1405-1416. doi: 10.1016/S0140-6736(13)60222-6. Epub 2013 Apr 12. PMID 23582727
- [Background] Ahs JW, Tao W, Löfgren J, Forsberg BC. Diarrheal diseases in low-and middle-income countries: incidence, prevention, and management. Open Infect Dis J. 2010; 4(1):113-24.
- [Background] Crider KS, Yang TP, Berry RJ, Bailey LB. Folate and DNA methylation: a review of molecular mechanisms and the evidence for folate's role. Adv Nutr. 2012 Jan;3(1):21-38. doi: 10.3945/an.111.000992. Epub 2012 Jan 5. PMID 22332098
- [Background] Kadhum RJ, Alghizzi EJ. The effect of oral folic acid supplementation on the course of acute infantile diarrhea. J Kerbala Univ. 2010; 8(4):177-82.
- [Background] Amelia A, Sinohaji AB, Supriatmo. Folic acid and acute diarrhea in children. Pediatr Indones. 2014; 54(5):273-9
- [Background] Niederberger KE, Dahms I, Broschard TH, Boehni R, Moser R. Safety evaluation of calcium L-methylfolate. Toxicol Rep. 2019 Sep 26;6:1018-1030. doi: 10.1016/j.toxrep.2019.09.012. eCollection 2019. PMID 31673504